CLINICAL TRIAL: NCT06220708
Title: Effects Of Dance Movement Therapy On Compassionate Flow In Nursing Students: An Experimental Study
Brief Title: Effects Of Dance Movement Therapy On Compassionate Flow In Nursing Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mackay Medical College (Other)
Responsible Party: Principal Investigator, Chin-Tsung Shen, the Office of Research and Development, Mackay Medical College
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: MMC-RD-112-1B-P001
Record Dates: First submitted 2024-01-15; First posted 2024-01-24 (Actual); Last update posted 2024-05-01 (Actual); Status verified 2024-04

CONDITIONS: Compassion; Educational Problems; Competence
Keywords: Compassion; dance movement therapy; nursing competence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The intervention group (Experimental): The intervention group underwent dance movement therapy.
  Interventions: Other: dance movement therapy
- The control group (Other): The control group received yoga training.
  Interventions: Other: yoga training

INTERVENTIONS:
Other: dance movement therapy — Our DMT program was adapted from an integrated somatic dance and visual arts program previously applied to the older population (Hsu, 2023). The intervention was scheduled in the afternoon and lasted for approximately 2 h. As previously recommended, rhythmic and contralateral movements on both sides of the body were emphasized in this study to enhance coordination and stimulation between the left and right cerebral hemispheres (Phillips-Silver and Trainor, 2007). The experimental groups were then subdivided into six groups. Balloons half-filled with water were used as the game in this study to guide individual and grouping rhythms and movements. Additionally, painting was incorporated to help participants understand their bodies and psychological states (Tjasink et al., 2023). Finally, group discussions and mutual support, along with verbal sharing after the DMT exercise, were encouraged.
  Arms: The intervention group
Other: yoga training — The yoga program included breathing exercises, Asanas, eye focus, body lock, and meditation. Participants were instructed to adjust their positioning based on their skill level to mitigate the risk of injury. The yoga intervention was scheduled at 2 pm and lasted for approximately 2 h.
  Arms: The control group

SUMMARY:
This study aimed to investigate the differences in compassionate flow among nursing students both before and after an educational intervention.

DETAILED DESCRIPTION:
Background: Only a few studies have explored how compassion is taught to nursing students.

Aim: This study aimed to investigate the differences in compassionate flow among nursing students both before and after an educational intervention.

Design: This study employed a cluster randomised controlled trial design. Settings: This study was conducted in medical schools in Taiwan. Participants: We enrolled first- and second-year nursing students. Methods: The intervention group underwent dance movement therapy, while the control group received yoga training. Compassionate flow was assessed using the Compassionate Engagement and Action Scale and the Fears of Compassion Scale.

ELIGIBILITY:
Inclusion Criteria:

* Freshmen or sophomore nursing students
* Those taking a course in Complementary and Alternative Therapies
* Willingness to participate and agreeing to complete the questionnaire

Exclusion Criteria:

* Deafness
* Limb disorders

Ages: 19 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 59 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Compassionate Engagement and Action Scales | 1 week
  The Compassionate Engagement and Action Scales, developed by Gilbert et al. (2017), comprises three subscales assessing different aspects of compassion: compassion for self, compassion for others, and compassion from others, each consisting of 13 items.

SECONDARY OUTCOMES:
Fear of Compassion Scales | 1 week
  The Fear of Compassion Scales consist of three subscales designed to assess the fear of compassion: fear of compassion for others (10 items), fear of compassion from others (13 items), and fear of compassion for oneself (15 items) .

CONTACTS AND LOCATIONS:
Overall Officials: Sheng-Miauh Huang, PhD, Principal Investigator — Department of Nursing, Mackay Medical College
Locations (1):
- Department of Nursing, New Taipei City, Taiwan

IPD SHARING:
Plan to Share IPD: No